CLINICAL TRIAL: NCT01738204
Title: The Women's Health Study: From Adolescence to Adulthood Sponsored by the Boston Center for Endometriosis.
Brief Title: The Women's Health Study: From Adolescence to Adulthood
Acronym: WHS:A2A
Status: Active, not recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Marc R Laufer, Chief, Division of Gynecology, Boston Children's Hospital
Other Study IDs: IRB-P00004267
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Pain; Endometriosis; Dysmenorrhea; Infertility
Keywords: endometriosis; dysmenorrhea; pelvic pain; women's health; adolescence; biorepository; observational; women; female; gynecology; fertility; infertility
MeSH Terms: conditions — Pelvic Pain; Endometriosis; Dysmenorrhea; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, saliva, blood, tissue, peritoneal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Females with endometriosis: Females with a surgical diagnosis of endometriosis or who undergoing surgery for suspected endometriosis. At this time, we are only recruiting patients of Boston Children's Hospital and Brigham and Women's Hospital for this group.
- Females without surgical diagnosis of endometriosis: Females do not need to be patients of Boston Children's Hospital or Brigham and Women's Hospital.

SUMMARY:
In order to learn more about women's health issues that occur over the lifespan, the Women's Health Study: from Adolescence to Adulthood is building a biorepository and database. The biorepository collects, processes and stores samples (such as urine, saliva, blood, cells, tissue and peritoneal fluid) until they are needed for research. The database contains de-identified information about our study participants. The biorepository and database are being created to serve as a resource for researchers from Boston Children's Hospital, Brigham and Women's Hospital and outside institutions.

ELIGIBILITY:
Inclusion Criteria:

* female
* at least 7 years old
* not experiencing natural menopause

Exclusion Criteria:

-

Ages: 7 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: clinic and community sample
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-11; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Establishing a biorepository and database | next 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc R Laufer, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

REFERENCES:
- See also: Women's Health Study: From Adolescence to Adulthood homepage — http://www.whsboston.org